CLINICAL TRIAL: NCT02571868
Title: Acute and Cronic Evaluation of AV/PV and VV Delay IEGM Based Optimisation Algorithm (QuickOpt™) Compared With Echocardiographic Method for Cardiac Resincronization Therapy in CRT Implants With Right Interventricular Basal-Mid Septum Placement of Leads (QuickSept Study)
Brief Title: Acute and Cronic Evaluation of AV/PV and VV Delay IEGM Based Optimisation Algorithm-QuickSept Study
Acronym: QuickSept
Status: Completed | Type: Observational
Sponsor: Maria Vittoria Hospital (Other)
Responsible Party: Principal Investigator, Dr.Massimo Giammaria, MD, Maria Vittoria Hospital
Other Study IDs: 002
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Optimization CRT-D

SUMMARY:
AtrioVentricular (AV) and InterVentricular (VV) delay optimization can improve ventricular function in Cardiac Resynchronization Therapy (CRT) and is usually performed by means of echocardiography. St Jude Medical has developed an automated algorhythm which calculates the optimal AV and VV delays (QuickOptTM) based on Intracardiac ElectroGrams, (IEGM), within 2 minutes. So far, the efficacy of the algorhythm has been tested acutely with standard lead position at right ventricular (RV) apex. Aim of this project is to evaluate the algorhythm performance in the mid- and long-term with RV lead located in mid-septum.

DETAILED DESCRIPTION:
Primary end-point was to evaluate the relationship between the series of aortic flow Velocity Time Integral (aVTI) values calculated by the two methods at the PV, AV, and VV interval settings recommended by both the QuickOptTM and the standard ECHO optimization in CRT-D patients, at three index times: pre-discharge, at 6-month and at 12-month follow-ups.

Secondary end-point was to define the correlation between the optimal AV, PV and VV intervals defined by ECHO, using aVTI measurements and by the QuickOptTM algorithm, IEGM-based.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CRT-D
* stable and safe placement of an active-fixation RV lead on mid-interventricular septum;
* achievement of an efficacious LV intravenous pacing from a Coronary Sinus (CS) branch.

Exclusion Criteria:

* AF
* Patients without spontaneous rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CRT-D
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Correlation between QuickOptTM and standard ECHO optimization | 12-month
  The primary endpoint was assessed by means the linear correlation analysis by the Pearson product-moment correlation coefficient to assess the agreement between the ECHO-based and the IEGM-based aVTIs for each of the AV/PV, and VV delay determinations

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Maria Vittoria, Torino, Italy, Italy